CLINICAL TRIAL: NCT06555523
Title: Comparison of Trigger Point Injection Application Methods in Patients With Fibromyalgia Syndrome and Myofascial Pain Syndrome
Brief Title: Trigger Point Injection in Patients With Myofascial Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Firat University (Other)
Responsible Party: Principal Investigator, Songül Bağlan Yentür, Firat University, Firat University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024/03-10
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2024-08-15 (Actual); Status verified 2024-08

CONDITIONS: Injection Site; Fibromyalgia
Keywords: Myofascial pain syndrome; Injection; Trigger point
MeSH Terms: conditions — Fibromyalgia; Myofascial Pain Syndromes

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided injection (Experimental): The skin will be cleaned with a suitable antiseptic solution and a sterile, 25 G, 1.5 inch dental-tipped needle will be used. Patients will be injected with 5 ml 2% lidocaine + 5 ml 0.9% NaCl. The linear probe (PLT-704SBT, 7.5 MHz) of the ultrasound device will be kept parallel to the trapezoidal fibers on the marked trigger point and the dental-tipped needle will be directed to the targeted point in plane with real-time imaging
  Interventions: Other: Ultrasound guided injection
- Blinded injection (Experimental): The skin will be cleaned with a suitable antiseptic solution and a sterile, 25 G, 1.5 inch dental-tipped needle will be used. Patients will be injected with 5 ml 2% lidocaine + 5 ml 0.9% NaCl. The needle will be directed to the most sensitive point and advanced until it will be reached the trigger point.
  Interventions: Other: Blinded injection

INTERVENTIONS:
Other: Ultrasound guided injection — The skin will be cleaned with a suitable antiseptic solution and a sterile, 25 G, 1.5 inch dental-tipped needle will be used. Patients will be injected with 5 ml 2% lidocaine + 5 ml 0.9% NaCl. The linear probe (PLT-704SBT, 7.5 MHz) of the ultrasound device will be kept parallel to the trapezoidal fibers on the marked trigger point and the dental-tipped needle will be directed to the targeted point in plane with real-time imaging
  Arms: Ultrasound-guided injection
Other: Blinded injection — The skin will be cleaned with a suitable antiseptic solution and a sterile, 25 G, 1.5 inch dental-tipped needle will be used. Patients will be injected with 5 ml 2% lidocaine + 5 ml 0.9% NaCl. The needle will be directed to the most sensitive point and advanced until it will be reached the trigger point.
  Arms: Blinded injection

SUMMARY:
This study aims to compare the effectiveness of blinded versus ultrasound-guided trigger point injections into the trapezius muscle in patients with FMS. Seventy-five patients with FMS will participate in this study. They will be randomly assigned to one of two groups: one group received ultrasound-guided trigger point injections, while the other group received blinded trigger point injections. Both groups will follow the same home exercise regimen, which included stretching and posture exercises targeting the trapezius and pectoral muscles. The effectiveness of the treatments was evaluated one month post-treatment. The assessment tools will include the Fibromyalgia Impact Questionnaire (FIQ) for function, the Visual Analog Scale (VAS) for pain, the Beck Anxiety Inventory (Beck-A) for anxiety, and the Neck Disability Questionnaire (NDQ) for neck disability.

DETAILED DESCRIPTION:
The primary objectives in treating Fibromyalgia Syndrome (FMS) are to deactivate trigger points, alleviate pain, and remove factors that exacerbate the condition. Recently, the use of ultrasound (US) has been advocated to reduce potential complications during trigger point injections and to ensure more effective administration of the treatment.This study aims to compare the effectiveness of blinded versus ultrasound-guided trigger point injections into the trapezius muscle in patients with FMS. Seventy-five patients with FMS will participate in this study. They will be randomly assigned to one of two groups: one group received ultrasound-guided trigger point injections, while the other group received blinded trigger point injections. Both groups will follow the same home exercise regimen, which included stretching and posture exercises targeting the trapezius and pectoral muscles. The effectiveness of the treatments was evaluated one month post-treatment. The assessment tools will include the Fibromyalgia Impact Questionnaire (FIQ) for function, the Visual Analog Scale (VAS) for pain, the Beck Anxiety Inventory (Beck-A) for anxiety, and the Neck Disability Questionnaire (NDQ) for neck disability.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 20-60 years who met the 2013 ACR criteria
* Patients who will be diagnosed with FMS and cervical chronic MAS according to Travel and Simons' criteria
* Patients who had a palpated tense band in the upper trapezius muscle and at least 1 active trigger point

Exclusion Criteria:

* Patients with a diagnosis of cervical radiculopathy, myelopathy, local or systemic infection, treatment for MAS in the last 3 months
* Patients who have symptom duration less than 3 months
* Patients with pregnancy status, acute or chronic disease that would cause clinical confusion at the time of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-09-20 (Estimated); Study Completion 2024-09-20 (Estimated)

PRIMARY OUTCOMES:
Pain assessment | 1 minute
  The pain levels of the patients in the last week will be questioned using a 0-10 cm long Visual Analog Scale (VAS). "0" indicated that the patient have no pain and "10" indicated that the patient's pain is unbearably severe

SECONDARY OUTCOMES:
Neck disability assessment | 2 minutes
  Neck Disability Questionnaire will be used. It consists of 10 questions questioning the effect of neck pain on pain sensitivity, personal care, weight lifting, reading, headaches, concentration, work/study, driving, sleep and social activities.
Functional assessment | 2 minutes
  Fibromyalgia Impact Questionnaire will be used. The FIQ is a 10-item scale that evaluates the health status and physical function of patients with fibromyalgia syndrome.

CONTACTS AND LOCATIONS:
Locations (1):
- Songul, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No